CLINICAL TRIAL: NCT00263432
Title: Reparation of Cartilage Injuries in the Human Knee by Implantation of Fresh Human Allogenic Chondrocytes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001/245
Record Dates: First submitted 2005-12-04; First posted 2005-12-08 (Estimated); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Cartilage Injuries in the Human Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Implantation of fresh human allogenic chondrocytes
  Interventions: Procedure: Human allogenic chondrocytes

INTERVENTIONS:
Procedure: Human allogenic chondrocytes — Implantation of fresh human allogenic chondrocytes in human knee cartilage injuries

SUMMARY:
Implantation of fresh human allogenic chondrocytes in human knee cartilage injuries to obtain a repair and prevention of secondary osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Important cartilage injury in the knee

Exclusion Criteria:

* Important axis deviation
* Inflammatory joint disorder
* Severe obesity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Healing of the cartilage injuries | After 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karl Fredrik Almqvist, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be